CLINICAL TRIAL: NCT01749306
Title: A Multicenter, Prospective, Randomized, Open-label, Intra-subject Controlled Study of the Efficacy and Safety of ABH001 for the Treatment of Stalled Chronic Cutaneous Wounds Associated With Generalized Epidermolysis Bullosa
Brief Title: A Study of the Efficacy and Safety of ABH001 in the Treatment of Patients With Epidermolysis Bullosa Who Have Wounds That Are Not Healing
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Shire Regenerative Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EB01-ABH001; 2012-001815-21 (EudraCT Number)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Epidermolysis Bullosa
Keywords: epidermolysis bullosa, chronic wound, wound healing, dermal repair, fibroblasts, Dermagraft
MeSH Terms: conditions — Epidermolysis Bullosa

ARMS (2):
- ABH001 (Other): ABH001 application plus wound care dressings.
  Interventions: Biological: ABH001
- Control (Other): Control wound treatment
  Interventions: Other: Control wound treatment

INTERVENTIONS:
Biological: ABH001 — ABH001 applications topically every 4 weeks (±1 week) with protocol-specified dressings until wound healed or up to 44 weeks
  Other Names: Dermagraft, Allogenic Neonatal Dermal Fibroblasts Seeded on poly(glycolide-co-L-lactide) (PGLLA) Scaffold
  Arms: ABH001
Other: Control wound treatment — Control wound care with protocol-specified dressings every 4 weeks (±1 week) up to 20 weeks with optional cross-over to ABH001 for additional 20 weeks
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ABH001 in the treatment of patients with epidermolysis bullosa who have wounds that are not healing.

It is hypothesized that ABH001 may initiate and continue wound healing in patients with epidermolysis bullosa.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal guardian must have read, understood and signed an Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent or Assent Form and must be able to and willing to follow study procedures and instructions
2. Male and female subjects.
3. Stable nutritional status.
4. Subjects with a confirmed diagnosis of generalized Epidermolysis Bullosa (EB)
5. Cutaneous wounds meeting the following criteria:

   1. Anatomical location: arms, legs, thorax, or back above the waistline and below the neck.
   2. Documented age (duration) of the wound(s).
   3. One or more wounds capable of potentially meeting the following wound selection criteria at the end of the observation period:

   i. Two clinically non-infected cutaneous wounds with no clinically meaningful change in wound size during the observation period.

   ii. Two matched wounds.
6. Negative urine pregnancy test for women of child-bearing potential.
7. Female subjects of childbearing potential and male subjects of procreative capacity must agree to use an effective method of contraception.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Diagnosis of non-genetic generalized EB.
3. Localized, active clinical infection of study wounds.
4. Diseases or conditions that could interfere with the assessment of safety and efficacy of the study treatment and compliance of the subject with study visits/procedures.
5. Known allergy to bovine products.
6. Known allergy to silver products.
7. Systemic infection at the time of enrolment in the study.
8. Currently receiving or have received oral steroid therapy within the previous 4 weeks.
9. Taking, or have participated in other clinical studies involving gene therapy, stem cell therapy, recombinant DNA/protein therapy.
10. Received ABH001, or other biologic or cell therapy for the treatment of EB in the study wound sites within the previous 3 months.
11. Hypersensitivity to any of the therapeutic agents.
12. History of malignant skin disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in wound surface area | 24 weeks

SECONDARY OUTCOMES:
Change in wound pain and wound itch | 24 weeks
Patient global impression of change (PGIC) | 24 weeks
Clinician global impression of change (CGIC) | 24 weeks
Proportion of subjects achieving reduction in wound surface area | 24 weeks
Time to reduction of wound surface area and duration of reduction | 24 weeks
Durability of wound healing | 24 weeks
Incidence, relatedness and severity of adverse events | Up to 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Arbuckle, MD, FAAD, FAAP, Principal Investigator — H&E Enterprises
Locations (14):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Lucile Packard Children's Hospital at Stanford University, Redwood City, California
  - Rady Children's Hospital - San Diego/UCSD, Pediatric and Adolescent Dermatology, San Diego, California
  - Denver Children's Hospital, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Virginia Clinical Research, Inc, Norfolk, Virginia
- Landeskrankenhaus Salzburg-Universitätsklinikum der Paracelsus Medizinischen Privatuniversität, Salzburg, Salzburg, Austria
- Canada (2):
  - Toronto Regional Wound Healing Clinic, Mississauga, Ontario
  - University of Montreal, Montreal, Quebec
- Hôpital Necker-Enfants Malades, Paris, Île-de-France Region, France
- University of Freiburg (Studiensekretariat Hautklinik Universitätsklinikum Freiburg - Hautklinik), Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Warszawki Uniwersytet Medyczny Katedra I Klinika Dermatologiczna, Warsaw, Masovian Voivodeship, Poland
- Hospital CUF Descobertas, Lisbon, Lisbon District, Portugal
- Hospital Universitario La Paz, Madrid, Madrid, Spain